CLINICAL TRIAL: NCT06981481
Title: Post-marketing Clinical Monitoring of Safety and Performance of the Silimed® Brand Breast Tissue Expander for Breast Reconstruction
Brief Title: Post-marketing Clinical Monitoring of Safety and Performance of Breast Tissue Expander for Breast Reconstruction
Acronym: STEPS-R
Status: Not yet recruiting | Type: Observational
Sponsor: Silimed Industria de Implantes Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: 70020
Record Dates: First submitted 2025-04-25; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Safety and Performance; Breast Tissue Expander
Keywords: post-market; safety; performance; Breast tissue expander; breast reconstruction
MeSH Terms: interventions — Tissue Expansion Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women undergoing breast reconstruction with Silimed® breast tissue expander.: Women undergoing breast reconstruction with Silimed® brand breast tissue expander since the elegibility criterea was attended.
  Interventions: Device: Breast tissue expander

INTERVENTIONS:
Device: Breast tissue expander — Silimed brand breast tissue expander

SUMMARY:
The study investigates the safety and performance of Silimed® brand breast tissue expander in women born with indication for breast reconstruction. The safety of the breast tissue expander will be evaluated by estimating known and unexpected adverse event rates through patient reports of adverse events after implantation. The performance of using Silimed® brand breast tissue expander will be evaluated by evaluating the assessment of tissue quality and satisfaction by the evaluating physician after implantation.

ELIGIBILITY:
Inclusion Criteria:

1. provide written informed consent
2. female sex at birth;
3. be 18 years of age or older;
4. have an indication for reconstruction with breast expander + breast implant(s);
5. have a plan to receive an expander with a textured surface from the Silimed® brand + implant breast with textured surface from the Silimed® brand;
6. ability to comply with the protocol throughout the follow-up period.

Exclusion Criteria:

1. breast augmentation without reconstruction in at least one breast;
2. neoplasia of any type (except breast neoplasia), not yet treated or under treatment, or requiring surgical removal at the time of implantation;
3. pregnancy or breastfeeding at the time of implantation;
4. smoking, uncontrolled diabetes, obesity (from grade 2) and ASA III/IV;
5. active infection not yet treated or being treated at any site at the time of implantation;
6. report or record of adverse reactions or intolerance to silicone prior to implantation;
7. immune diseases that affect connective tissue in activity or under treatment (e.g. lupus erythematosus, discoid lupus, scleroderma, etc.) at the time of implantation;
8. record or report of use of illicit drugs or medications that increase the risk of immediate post-surgical complications (eg, medications that interfere with coagulation);
9. high surgical risk or complications in the immediate post-surgery period, estimated before the implantation;
10. evidence or report of tissue characteristics that are clinically inconsistent with a successful implantation (eg tissues with excessive fibrosis or compromised vascularization);
11. may not have participated in another clinical study up to 6 months before placement of the expander, unless the researcher deems it to be good for the participant and not impact the study;
12. previous treatment with radiotherapy;
13. any other condition that, based on the opinion of the researcher or designee, may prevent the provision of informed consent, make study participation unsafe, compromise adherence to the protocol, complicate the interpretation of study outcome data or otherwise interfere with the achievement of the study objectives.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Born females with indication of breast reconstruction using Silimed brand breast tissue expander.
Sampling Method: Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through study completion, an average of 1 year
  Estimate adverse events rate for breast tissue expander
Evaluator's Satisfaction in Relation to expansion | Through study completion, an average of 1 year
  Estimate the performance of Silimed® brand breast tissue expander with through the satisfaction of the evaluator (investigator) regarding the result of the expansion so far. The assessment will be done by means of a likert scale, where the following satisfaction options can be selected: 1 = definitely unsatisfied, 2 = unsatisfied, 3 = slightly satisfied, 4 = satisfied and 5 = definitely satisfied.
Evaluator's Assessment of tissue quality | Through study completion, an average of 1 year
  The assessment of tissue quality is clinical and will occur at every visit, including the final assessment. Estimate the performance of Silimed® brand breast tissue expander with textured surface throught the satisfaction of the evaluator regarding the vascularization, innervation, color and texture of and quality of the expanded tissue.
  To measure satisfaction, a Likert scale where the following satisfaction options can be marked: 1 = definitely dissatisfied, 2 = dissatisfied, 3 = somewhat satisfied, 4 = satisfied and 5 = definitely satisfied.
  Satisfaction will be measured in percentages of each category of the Likert scale in each follow-up time. Values from 0 to 20 will be considered poor results, bad results from 21 to 40, intermediate results from 41 to 60, good results from 61 to 80, and excellent results from 81 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo A Bello, Principal Investigator — Hospital de câncer - HCIII (INCA)
Locations (2):
- Brazil (2):
  - Hospital de câncer HCIII (INCA), Rio de Janeiro, Rio de Janeiro
  - Fundação do ABC - Centro universitário FMABC, Santo André, São Paulo